CLINICAL TRIAL: NCT06951100
Title: Mechanisms of Myocardial Injury and Ischemia in Patients With Rapid Atrial Fibrillation
Acronym: Mi-AF
Status: Recruiting | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: British Heart Foundation (Other); NHS Lothian (Other Government)
Responsible Party: Sponsor
Other Study IDs: AC24081; 25-SS-0009 (Other: Health Research Authority (HRA))
Record Dates: First submitted 2025-04-28; First posted 2025-04-30 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-04

CONDITIONS: Atrial Fibrillation (AF)
Keywords: Atrial Fibrillation; Cardiology; Emergency Medicine; Myocardial Infarction; Myocardial Ischemia; Coronary Artery Disease
MeSH Terms: conditions — Atrial Fibrillation; Myocardial Infarction; Myocardial Ischemia; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples (plasma and serum)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CT coronary angiography — To assess the presence of obstructive coronary artery disease, participants will either have coronary angiography as part of their routine care or they will return for a research CT scan of their heart (CT Coronary Angiogram)

SUMMARY:
The goal of this observational study is to better understand the role of measuring troponin (a protein measured by a blood test) and coronary imaging in patients presenting with rapid atrial fibrillation (AF)

The main questions this study aims to answer are:

1. Are patients with a fast, irregular heartbeat (rapid AF) and damage to the heart (myocardial injury) more likely than those without damage to the heart to have blocked heart arteries (obstructive coronary artery disease)
2. Are patients with a fast, irregular heartbeat (rapid AF) and damage to the heart (myocardial injury) with further evidence that their heart hasn't been getting enough oxygen (myocardial ischemia) more likely to have imaging evidence of myocardial infarction than those without myocardial ischemia

To do this, we will measure troponin in patients with rapid AF and then carry out further investigations of the heart (electrocardiogram, echocardiogram, CT scan and cardiac MRI)

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and over
2. Primary presentation with symptoms related to atrial fibrillation
3. Atrial fibrillation with a ventricular rate >100 bpm on a 12-lead electrocardiogram
4. Able to provide informed consent

Exclusion Criteria

1. Previous myocardial infarction
2. Previous coronary revascularisation procedure
3. Patients in renal failure (eGFR <30ml/min/1.73m2) or major allergy to contrast media
4. Pregnancy or breast feeding
5. Deemed unsuitable for participation in the study by the attending clinician
6. Previous enrolment in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to an Emergency Department or Acute Medical Unit with rapid atrial fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Presence of obstructive coronary artery disease | within 4 weeks of presentation
  Presence of obstructive coronary artery disease as defined as at least one stenosis ≥70% in a major epicardial coronary artery or ≥50% in the left main stem on CTCA or invasive coronary angiography

SECONDARY OUTCOMES:
Imaging evidence of new myocardial infarction | within 4 weeks of presentation
  Imaging evidence of new myocardial infarction

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, East of England, United Kingdom

IPD SHARING:
Plan to Share IPD: No